CLINICAL TRIAL: NCT01972360
Title: Non-isotope Based Imaging Modalities vs 99mTcSPECT to Detect Myocardial Ischemia in Patients at High Risk for Ischemic Cardiovascular Events
Brief Title: Non-isotope Based Imaging Modalities vs Technetium-99m Single-Photon Emission Computed Tomography(99mTcSPECT)
Acronym: MITNECB5
Status: Completed | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: MITNEC B5
Record Dates: First submitted 2013-07-18; First posted 2013-10-30 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Myocardial Ischemia
Keywords: SPECT; CMR; High risk for ischemic cardiovascular events
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Diagnosis: Group 3: 99mTCSPECT plus stress echocardiography
- group 1 : diagnosis: Group 1: 99mTcSPECT plus CMR
- Group 2: diagnosis: Group 2: 99mTcSPECT plus CT

SUMMARY:
SPECT is currently the dominant clinical test for diagnostic and prognostic purposes as well as therapeutic decision-making. Given the shortage of nuclear reactor-produced Tc, advancing the use of non-isotope based imaging modalities has the potential to change the standard of care for patients with CAD as each one of these technics (CMR, CT, Stress echocardiography) has its own distinct potential advantages over SPECT.

DETAILED DESCRIPTION:
Obtain a better understanding of the clinical utility of advanced non-isotope-based imaging modalities to detect relevant CAD as potential alternatives to SPECT. Approximately 450 subjects will be enrolled in total. Three groups of about 150 patients per group. Each group will undergo imaging with 2 modalities; Group 1: 99mTcSPECT plus CMR, Group 2: 99mTcSPECT plus CT, Group 3:99mTcSPECT plus stress echocardiography. All 450 patients will undergo standard invasive coronary angiography following completion of non-invasive imaging, except for patients in whom both nuclear and non-nuclear imaging modalities reveal a normal result confirming the absence of significant coronary artery disease (i.e invasive angiography would not be clinically indicated and FFR would be considered to be above 0.8). Thrombolysis in Myocardial Infraction (TIMI) flow will be measured in all patients undergoing angiography, and fractional flow reserve (FFR) will be measured in all patients except those with TIMI flow =0, 1 and 2. All imaging procedures must be completed within 6 weeks. All patients will have a follow-up visit at 6 months after enrollment. During the 6 month follow-up visit major adverse cardiovascular events will be collected and adjudicated by a clinical endpoint committee (CEC).

ELIGIBILITY:
Inclusion Criteria:

* clinically indicated request for SPECT
* ability to undergo at least one of three non-nuclear imaging tests; CMR, CT or Stress Echocardiography
* History of recent symptoms suggestive of myocardial ischemia
* High risk for ischemic cardiovascular events

Exclusion Criteria:

* severely reduced systolic function (LV ejection fraction less than 35%)
* Recent (less than 3 days) acute coronary syndrome including acute myocardial infarction
* contraindications to dipyridamole SPECT including : i)severe reactive airway disease; ii) less than 3 days post Myocardial Infarction - Acute Coronary Syndrome (MI-ACS); iii) high-grade Atrioventricular block (AV block); iv)allergy to dipyridamole or theophylline; v) caffeine within 12 hours; vi) theophylline use within 48 hours; vii) severe claustrophobia; or viii) women who may be pregnant
* kidney dysfunction (i.e estimated Glomerular Filtration Rate (eGFR) less than 45)
* use of investigational drug or device within 30 days of screening visit
* Coronary Artery Bypass Graft(s) surgery (CABG)

Ages: 18 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 450 patients across Canada. Patients will be identified after a clinically indicated SPECT for evaluation of myocardial ischemia.The investigator will assign the patient in one of the three groups based on his medical assessment and availability of equipment at the centre.
Sampling Method: Non-Probability Sample
Enrollment: 467 (Actual)
Dates: Start 2012-10; Primary Completion 2018-05 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
Overall accuracy of "significant coronary artery disease (CAD)" according to non-invasive imaging modality | baseline
  The overall accuracy is calculated as the probability that a subject is correctly classified (presence of significant CAD or not) by non-invasive imaging modality. The standard of truth is presence of significant CAD or not according to the invasive fractional flow reserve (FFR)
Sensitivity of "significant CAD" according to non-invasive imaging modality | baseline
  The sensitivity is calculated as the probability that a subject with presence of significant CAD according to FFR is correctly identified as such by non-invasive imaging modality
Specificity of "significant CAD" according to non-invasive imaging modality | baseline
  The specificity is calculated as the probability that a subject with absence of significant CAD according to FFR is correctly identified as such by non-invasive imaging modality
Positive predictive value of "significant CAD" according to non-invasive imaging modality | baseline
  The positive predictive value is calculated as the probability that a subject with presence of significant CAD according to non-invasive imaging modality truly have significant CAD according to FFR
Negative predictive value of "significant CAD" according to non-invasive imaging modality | Baseline
  The negative predictive value is calculated as the probability that a subject with absence of significant CAD according to non-invasive imaging modality truly does not have significant CAD according to FFR

SECONDARY OUTCOMES:
Overall accuracy of "high-risk CAD" according to non-invasive imaging modality flow and FFR | baseline
Sensitivity of "high-risk CAD" according to non-invasive imaging modality flow and FFR | Baseline

OTHER OUTCOMES:
Specificity of "high-risk CAD" according to non-invasive imaging modality flow and FFR | baseline
Positive predictive value of "high-risk CAD" according to non-invasive imaging modality flow and FFR | baseline
Negative predictive value of "high-risk CAD" according to non-invasive imaging modality flow and FFR | baseline
Overall accuracy of "high-risk CAD" according to non-invasive imaging modality to predict occurrence of the composite clinical endpoint of major adverse cardiovascular events (MACE) | baseline
Sensitivity of "high-risk CAD" according to non-invasive imaging modality to predict occurrence of the composite clinical endpoint of major adverse cardiovascular events (MACE) | baseline
Specificity of "high-risk CAD" according to non-invasive imaging modality to predict occurrence of the composite clinical endpoint of major adverse cardiovascular events (MACE) | baseline
Positive predictive value of "high-risk CAD" according to non-invasive imaging modality to predict occurrence of the composite clinical endpoint of major adverse cardiovascular events (MACE) | baseline
Negative predictive value of "high-risk CAD" according to non-invasive imaging modality to predict occurrence of the composite clinical endpoint of major adverse cardiovascular events (MACE) | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Tardif, M.D, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided